CLINICAL TRIAL: NCT06492798
Title: Effectiveness and Safety of Mesenchymal Stem Cell Therapy in Long COVID Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Dong Yuchao, Professor., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSCinLong-COVID
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Long COVID; Post-Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; Mesenchymal stem cell; Effectiveness; Safety
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants will receive intravenous infusion of MSCs once or an additional infusion on days 35-42.
  Dosage: 1×10^6 cells per kilogram of body weight Specification: 1×10^7 cells/100ml
  Interventions: Drug: umbilical cord mesenchymal stem cell
- Placebo group (Placebo Comparator): Participants will receive intravenous infusion of placebo Dosage: 10ml per kilogram of body weight
  Interventions: Drug: umbilical cord mesenchymal stem cell

INTERVENTIONS:
Drug: umbilical cord mesenchymal stem cell — intravenous infusion of umbilical cord mesenchymal stem cell
  Other Names: MSCs

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of mesenchymal stem cell therapy in long-COVID patients. The main questions it aims to answer include:

* whether umbilical cord mesenchymal stem cell therapy does benefit long-COVID patients
* whether umbilical cord mesenchymal stem cell therapy is safe for long-COVID patients.

Participants' demographics, chief complaints, and vital signs will be collected and recorded. Basic physical examinations, bloodwork routine, biochemical indexes, oxygen saturation (SpO2) levels, 6-minute walk tests, high-resolution computed tomography (HRCT) scan (if necessary) results will be conducted.

Participants will receive either an intravenous infusion of mesenchymal stem cells, or a placebo for one time. Participants' symptoms will be assessed on Day 28 of the trial. If there is no significant effect, an additional infusion will be given on Days 35-42, and the symptoms will be reassessed 28 days after that.

Continuous nebulized inhalation of UCMSC-derived exosomes will be administered for 5 days twice daily to treatment group, with no treatment given to the control group. Researchers will compare data and information collected from the treatment and control groups to evaluate the safety and efficacy of UCMSC-derived exosomes for the treatment of chronic cough after COVID-19 infection.

DETAILED DESCRIPTION:
Since the outbreak of the COVID-19 pandemic, according to the official statistics from the WHO website, there have been over 694 million confirmed cases worldwide until August 2023, with approximately 6.9 million deaths. In addition to the high incidence and mortality rates in the initial weeks following infection, up to 70% of COVID-19 patients may experience long-term complications, significantly impacting human health and placing a substantial burden on hospital resources.

A study evaluated 2,320 adult participants who were discharged between March 7, 2020, and April 18, 2021 from several National Health Service (NHS) hospitals in the United Kingdom, and found that only 25.5% of COVID-19 patients had fully recovered five months after discharge. And the improvement in patients' conditions was minimal even when study period was extended to one year. 71% of patients continued to experience one or more post-COVID-19 sequelae, with common symptoms including fatigue, difficulty breathing, muscle pain, and insomnia, etc. According to multiple studies, post-COVID-19 sequelae may involve 203 different symptoms and affect 10 organ systems in the body, including the neurological, reproductive, cardiovascular, and pulmonary systems. The World Health Organization (WHO) published an official definition of long COVID in October 2021. They define it as a condition that "occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis." Despite some guidelines for the management of long COVID, there is still a lack of specific treatment methods. Currently, the most important strategy is vaccination. Vaccination can help alleviate symptoms during the acute infection period, and studies have found that individuals who are vaccinated against COVID-19 have approximately a 50% lower risk of developing long COVID compared to those who are unvaccinated. Also, there are other therapies that are in the clinical research stage, and one of which is stem cell therapy. Mesenchymal stem cells (MSCs) are a type of cell with self-renewal and multi-directional differentiation abilities. They are the primitive "seed cells" that form various tissues and organs in the human body. Under specific conditions, MSCs can differentiate into various cells in the human body, including osteoblasts, adipocytes, chondrocytes, and other cells of the stromal lineage, and repair tissue damage through the secretion of corresponding factors. Meanwhile, MSCs also act as "inflammation terminators" by regulating immune reactions through paracrine functions and interactions with immune cells. This ultimately leads to the downregulation of local inflammatory responses and alleviation of excessive immune reactions.

The research team led by Wang Fusheng published a study in the journal "eBioMedicine" (impact factor: 8.143) in 2022, which explored the use of umbilical cord mesenchymal stem cells (UC-MSCs) for the treatment of severe COVID-19 patients and followed up patients for one year. The study confirmed that UC-MSCs therapy, as an adjuvant therapy, has long-term benefits for lung injury in severe COVID-19 patients. This was a randomized, double-blind, controlled trial, with 100 patients randomly assigned in a 2:1 ratio (65 in the UC-MSCs group and 35 in the control group). The results showed that UC-MSCs helped in the resolution of lung consolidative lesions, with 17.9% of patients in the UC-MSCs group having normal CT images after one year of follow-up. In contrast, the control placebo group had not recovered from lung injury. There were no significant differences in the incidence of adverse events between the two groups. And in Japan, the Japanese Respiratory Syndrome Society has been conducting research on the long-term effects of COVID-19 since August 1, 2020. According to foreign media reports, the Kyushu Regenerative Medicine Special Committee in Japan has approved a program for the use of autologous adipose-derived mesenchymal stem cells in the treatment of post-COVID-19 syndrome. This patented technology developed by the Korean Stem Cell Research Institute has undergone a 120-day review and three rounds of screening by a committee of 16 experts from various fields, and has passed the review of the current regenerative medical plan for post-COVID-19 syndrome. The director of the Stem Cell Research Institute, who developed this therapy, stated, "This approval has received strong support from the Regenerative Medicine Special Committee. The investigators believe that mesenchymal stem cells, through their anti-inflammatory and tissue regeneration effects, will have good results in treating post-COVID-19 syndrome." This study aims to evaluate the effectiveness and safety of mesenchymal cell therapy for long COVID-19 patients. It is a prospective exploratory study, randomized, double-blind, placebo-controlled trial, planning to include a total of 76 patients who have been infected with COVID-19. By assessing the improvement of CTCAE 5.0 symptom scores in the treatment group and control group at 28 days, 12 weeks, and 24 weeks after treatment completion, the effectiveness and safety of mesenchymal stem cells in patients with long- term COVID-19 will be evaluated. This study is divided into two stages. Stage one: 10 patients will be enrolled, all receiving mesenchymal stem cell treatment, primarily assessing their safety. Stage two: 66 patients will be enrolled, randomly assigned in a 1:1 ratio to the treatment group and control group, evaluating the effectiveness and safety of mesenchymal stem cell therapy for long-term COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for Long COVID according to WHO.
* Main symptoms assessed based on CTCAE 5.0.
* Symptoms evaluated for exclusion reasons of other diseases by relevant specialists.
* No recent plans for pregnancy (negative pregnancy test within 72 hours for women of childbearing age prior to the start of the trial), and willing to use effective non-pharmaceutical contraceptive measures during the study.
* Signed informed consent forms and agreements to participate in this clinical trial.

Exclusion Criteria:

* Active malignant tumors.
* Active infections.
* Abnormal liver or kidney function (ALT, AST > 2 times the upper limit of normal; Cr > 2 times the upper limit of normal).
* Women who are pregnant, lactating, or planning to become pregnant during the trial.
* Participated in other clinical trials within the last 3 months prior to screening.
* Other reasons deemed inappropriate for participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Common Terminology Criteria for Adverse Events (CTCAE5.0) | 28th day
  CTCAE is a descriptive terminology which can be used for Adverse Event (AE) reporting. An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Higher grades mean worse outcome.

SECONDARY OUTCOMES:
Common Terminology Criteria for Adverse Events (CTCAE5.0) | 12th week, 24th week
  CTCAE is a descriptive terminology which can be used for Adverse Event (AE) reporting. An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Higher grades mean worse outcome.

OTHER OUTCOMES:
C reactive protein(CRP) | 28th day, 12th week, 24th week
  For paticipants with high C reactive protein level at enrollment, C reactive protein will be tested. Level of CRP change and time for its relief will be recorded.
Dosage of corticosteroids | 28th day, 12th week, 24th week
  For paticipants using corticosteroids to treat long COVID, total dosage and course of corticosteroids will be recorded.
SpO2 | 28th day, 12th week, 24th week
  For paticipants with pulmonary fibrosis, SpO2 will be tested and evaluated.
6-minute walk test | 28th day, 12th week, 24th week
  For paticipants with pulmonary fibrosis, 6-minute walk testwill be tested and evaluated.
HRCT scan | 28th day, 12th week, 24th week
  For paticipants with pulmonary fibrosis, HRCT scan will be tested and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchao Dong, Doctor, Study Director — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study information, including study protocol, statistical analysis plan, informed consent form, clinical study report will be available immediately upon the data being de-identified and properly revised for quality control on the study website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2-years
Access Criteria: The requested data will be shared with investigators via a secured, password-protected software website

REFERENCES:
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Ledford H. Can drugs reduce the risk of long COVID? What scientists know so far. Nature. 2022 Apr;604(7904):20-21. doi: 10.1038/d41586-022-00823-y. No abstract available. PMID 35338366
- [Background] Chen L, Qu J, Kalyani FS, Zhang Q, Fan L, Fang Y, Li Y, Xiang C. Mesenchymal stem cell-based treatments for COVID-19: status and future perspectives for clinical applications. Cell Mol Life Sci. 2022 Feb 20;79(3):142. doi: 10.1007/s00018-021-04096-y. PMID 35187617
- [Background] Yousefi Dehbidi M, Goodarzi N, Azhdari MH, Doroudian M. Mesenchymal stem cells and their derived exosomes to combat Covid-19. Rev Med Virol. 2022 Mar;32(2):e2281. doi: 10.1002/rmv.2281. Epub 2021 Aug 7. PMID 34363275
- [Background] Rebelatto CLK, Senegaglia AC, Franck CL, Daga DR, Shigunov P, Stimamiglio MA, Marsaro DB, Schaidt B, Micosky A, de Azambuja AP, Leitao CA, Petterle RR, Jamur VR, Vaz IM, Mallmann AP, Carraro Junior H, Ditzel E, Brofman PRS, Correa A. Safety and long-term improvement of mesenchymal stromal cell infusion in critically COVID-19 patients: a randomized clinical trial. Stem Cell Res Ther. 2022 Mar 21;13(1):122. doi: 10.1186/s13287-022-02796-1. PMID 35313959
- [Background] Zhao F, Ma Q, Yue Q, Chen H. SARS-CoV-2 Infection and Lung Regeneration. Clin Microbiol Rev. 2022 Apr 20;35(2):e0018821. doi: 10.1128/cmr.00188-21. Epub 2022 Feb 2. PMID 35107300
- [Background] Shi L, Wang L, Xu R, Zhang C, Xie Y, Liu K, Li T, Hu W, Zhen C, Wang FS. Mesenchymal stem cell therapy for severe COVID-19. Signal Transduct Target Ther. 2021 Sep 8;6(1):339. doi: 10.1038/s41392-021-00754-6. PMID 34497264
- [Background] Meng F, Xu R, Wang S, Xu Z, Zhang C, Li Y, Yang T, Shi L, Fu J, Jiang T, Huang L, Zhao P, Yuan X, Fan X, Zhang JY, Song J, Zhang D, Jiao Y, Liu L, Zhou C, Maeurer M, Zumla A, Shi M, Wang FS. Human umbilical cord-derived mesenchymal stem cell therapy in patients with COVID-19: a phase 1 clinical trial. Signal Transduct Target Ther. 2020 Aug 27;5(1):172. doi: 10.1038/s41392-020-00286-5. PMID 32855385
- [Background] Shi L, Yuan X, Yao W, Wang S, Zhang C, Zhang B, Song J, Huang L, Xu Z, Fu JL, Li Y, Xu R, Li TT, Dong J, Cai J, Li G, Xie Y, Shi M, Li Y, Zhang Y, Xie WF, Wang FS. Human mesenchymal stem cells treatment for severe COVID-19: 1-year follow-up results of a randomized, double-blind, placebo-controlled trial. EBioMedicine. 2022 Jan;75:103789. doi: 10.1016/j.ebiom.2021.103789. Epub 2021 Dec 25. PMID 34963099
- [Background] Shi L, Huang H, Lu X, Yan X, Jiang X, Xu R, Wang S, Zhang C, Yuan X, Xu Z, Huang L, Fu JL, Li Y, Zhang Y, Yao WQ, Liu T, Song J, Sun L, Yang F, Zhang X, Zhang B, Shi M, Meng F, Song Y, Yu Y, Wen J, Li Q, Mao Q, Maeurer M, Zumla A, Yao C, Xie WF, Wang FS. Effect of human umbilical cord-derived mesenchymal stem cells on lung damage in severe COVID-19 patients: a randomized, double-blind, placebo-controlled phase 2 trial. Signal Transduct Target Ther. 2021 Feb 10;6(1):58. doi: 10.1038/s41392-021-00488-5. PMID 33568628
- [Background] Zhou T, Yuan Z, Weng J, Pei D, Du X, He C, Lai P. Challenges and advances in clinical applications of mesenchymal stromal cells. J Hematol Oncol. 2021 Feb 12;14(1):24. doi: 10.1186/s13045-021-01037-x. PMID 33579329